CLINICAL TRIAL: NCT06609447
Title: A Multicenter Randomized, Double-blind, Placebo-controlled Study on the Efficacy and Safety of Combining Probiotic VSL#3 With Vedolizumab for the Treatment of Moderate Ulcerative Colitis
Brief Title: The Efficacy and Safety of Combining Probiotic VSL#3 With Vedolizumab for the Treatment of Moderate Ulcerative Colitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0602
Record Dates: First submitted 2024-09-22; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; Injections

STUDY DESIGN:
Intervention Model Description: A Multicenter, Randomized, Double-blind, Placebo-controlled trial in adult subjects with moderate active ulcerative colitis
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VSL#3 combine with Vedolizumab Arm (Experimental): Treatment with probiotic VSL#3 combined with vedolizumab; Subjects will receive two sachets daily of VSL#3, each containing 450 billion bacteria (totaling 900 billion bacteria per day), for 14 weeks.
  Vedolizumab will be administere as per clinical practice with the following schedule: 300 mg ev at 0, 2 and 6, 14 weeks.
  Interventions: Dietary Supplement: VSL#3; Drug: Vedolizumab
- Placebo combine with Vedolizumab Arm (Placebo Comparator): Treatment with placebo combined with vedolizumab; Subjects will receive two sachets daily of Placebo for 14 weeks. Vedolizumab will be administere as per clinical practice with the following schedule: 300 mg ev at 0, 2 and 6, 14 weeks.
  Interventions: Dietary Supplement: Placebo; Drug: Vedolizumab

INTERVENTIONS:
Dietary Supplement: VSL#3 — VSL#3 450 billion CFU/sachet
  Arms: VSL#3 combine with Vedolizumab Arm
Dietary Supplement: Placebo — Placebo sachets with maltose, cornstarch and dioxide
  Other Names: Placebo (for VSL#3)
  Arms: Placebo combine with Vedolizumab Arm
Drug: Vedolizumab — Patients will start combined therapy with vedolizumab and VSL#3 or placebo at the same time. Vedolizumab will be administered according to clinical practice with the following schedule: 300 mg intravenously on Baseline (Day 1 / Week 0) and Weeks 2, 6, and 14, with a flexibility of ±3 days relative to the start of VSL#3 administration.
  Other Names: Vedolizumab 300 mg Injection

SUMMARY:
An imbalance in the gut microbiota and mucosal immune dysfunction leading to intestinal inflammation are central to the pathogenesis of ulcerative colitis (UC). Both international and domestic inflammatory bowel disease (IBD) guidelines consistently recommend the use of the probiotic VSL#3 for inducing or maintaining remission in cases of mild-to-moderate UC. While the development of biologic therapies in recent years has provided new directions for IBD treatment, classic biologics such as infliximab may increase the risk of opportunistic infections and malignancies. Vedolizumab, when used for the induction therapy of UC, has a response rate of less than 80%, a slightly slower onset of action, and a slight increase in Clostridioides difficile infection (CDI) incidence. Currently, there is a lack of clinical data on the adjunctive use of VSL#3 with biologic agents in the treatment of UC globally.

Therefore, this project aims to design a multi-center, randomized, placebo-controlled, double-blind study. The primary objective is to compare the changes in clinical response in patients with moderately active UC treated with either VSL#3 or placebo in combination with vedolizumab (VDZ) for six weeks.

DETAILED DESCRIPTION:
This study enrolled patients aged 18-85 years with moderate ulcerative colitis and randomly assigned them in a 1:1 ratio to an experimental group and a control group. Patients in the experimental group received two packets of VSL#3 (450 billion CFU/packet) daily for 14 weeks, along with Vedolizumab (300 mg once weekly at weeks 0, 2, 6, and 14). The control group received placebo packets and Vedolizumab on the same schedule. The primary outcome was the proportion of patients with a decrease of ≥3 points in the SCCAI score at week 6, along with improvement in fecal calprotectin (FC) levels (decrease of ≥50% from baseline) at weeks 6 and 14. Secondary outcomes included clinical response, clinical remission, corticosteroid-free clinical remission, and changes in quality of life scores at week 14.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a man or woman aged 18-85 years, inclusive.
* Diagnosed with ulcerative colitis (UC) at least 90 days prior to baseline, supported by comprehensive colonoscopy findings and histopathological evidence obtained within the past year. Participants must provide full colonoscopy or sigmoidoscopy reports along with pathology results conducted within the last 3 months, as well as blood indicators (within 1 week) at baseline screening. Individuals currently experiencing infection, dysplasia, or malignancy will be excluded from participation.
* Subject has moderate active UC and had a Mayo score of 6-10 at screening.
* Planned treatment with Vedolizumab as initial therapy or reinduction, with reinduction defined as no vedolizumab treatment within 1 year.
* Confirmed by the investigator that despite receiving at least one of the following treatments, the subject has shown an inadequate response, loss of response, or intolerance:

  1. Oral aminosalicylates (e.g., mesalamine, sulfasalazine, olsalazine, balsalazide), where the subject exhibits ongoing signs and symptoms of active disease during at least 4 weeks of treatment with mesalamine 2.4 g/day, sulfasalazine 4 g/day, olsalazine 1 g/day, or balsalazide 6.75 g/day.
  2. Immunosuppressants: failure to respond after receiving at least 42 consecutive days of treatment with azathioprine, 6-mercaptopurine, or methotrexate (MTX) injections prior to baseline (Week 0), with minimum doses of azathioprine ≥ 0.75 mg/kg/day or 6-MP ≥ 0.5 mg/kg/day (rounded to the nearest tablet dose) or MTX ≥ 15 mg/week (SC/IM), or the highest tolerated dose due to adverse effects such as leukopenia, elevated liver enzymes, or nausea.
* No increase in dose of oral 5-ASA and Immunosuppressants could be allowed if it is maintained stable at least 2 weeks before screening.
* Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
* Willing and able to complete the required Subject Diary.
* Willing and able to meet all study requirements, including attending all assessment visits and phone calls.

Exclusion criteria:

* Diagnosis of Crohn's disease, undetermined IBD or other colitis.
* UC disease limited to the rectum (<15 cm from the anal verge)
* Steroid therapy initiation within 2 weeks before screening visit.
* Used antibiotics for intestinal or other infections within 2 weeks of the screening
* Use of other probiotics preparations within the last 2 weeks before study entry (screening)
* Used rectal 5-ASA within the past week before study entry (screening)
* Adjustment of oral 5-ASA and immunosuppressant dosages due to disease progression after colonoscopy screening until enrollment.
* Within 1 week prior to screening, the participant has taken nonsteroidal anti-inflammatory drugs (NSAIDs) or anti-diarrheal medications for 5 consecutive days.
* Positive Clostridioides difficile detection toxin results within the past month prior to screening.
* Pregnancy and breastfeeding women
* Other biologics/advanced therapies are used as concomitant therapy and Previous use of other biologics
* History of allergy to maltose and/or cornstarch and/or silica
* Subjects with severe primary heart, liver, lung, kidney, hematologic, or serious diseases that affect their survival, such as cancer, AIDS, asthma, kidney stones, renal dysfunction; urine protein >+, microscopic hematuria, ALT >2N (N is the upper limit of normal), Cr > normal upper limit, platelet count <50x10^9/L, white blood cell count <3.0x10^9/L.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-21 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Response rate at week 6 | At week 6
  The proportion of participants with a SCCAI score reduction of ≥3 points from baseline in the experimental group compared to the control group at week 6

SECONDARY OUTCOMES:
Clinical Response rate at week 14 | At Week 14
  The proportion of participants in the experimental group compared to the control group at week 14 with:
  * A reduction in modified Mayo score of ≥30% and ≥3 points from baseline, along with a decrease of ≥1 point in the rectal bleeding subscore or a subscore of 0 or 1.
  * Or a PRO2 score showing at least a 50% reduction in rectal bleeding and stool frequency.
  * Or a reduction in SCCAI score of ≥3 points.
Clinical Remission rate at week 14 | At Week 14
  The proportion of participants in the experimental group compared to the control group at week 14 with:
  * A modified Mayo score ≤2 points and no single item score >1 point.
  * Or a PRO2 score with a rating of 0 for rectal bleeding and stool frequency.
  * Or a SCCAI score ≤2 points.
Steroid-free Clinical Remission rate at week 14 | At Week 14
  The proportion of participants in the experimental group compared to the control group at week 14 with a modified Mayo score ≤2 points and no single item score >1 point, and who have completely tapered off steroids.
At week 2 on PRO2 and Urgency NRS through dairy daily | At Week 2
  At Week 2, assess the proportion of participants achieving a decrease in the PRO2 (Patient-Reported Outcome) scores for rectal bleeding and stool frequency, and the mean value of the Urgency Numeric Rating Scale (UNRS) for bowel movements.
Inflammatory Bowel Disease Questionnaire (IBDQ) variation | At the end of treatment weeks 6 and 14
  The difference between the IBDQ scores obtained at Week 14 and Week 6, compared to the baseline (initial) IBDQ scores taken before the start of the intervention or treatment.
The proportion of patients with a ≥50% decrease in fecal calprotectin (FC) and the changes in the Urgency Numeric Rating Scale (UNRS) | At the end of treatment weeks 6 and 14
  At Week 14 and Week 6, assess the proportion of participants achieving a decrease in fecal calprotectin (FC) levels of ≥50% from baseline, and the changes in the mean value of the Urgency Numeric Rating Scale (UNRS) from baseline.
Adverse Events | Through Week 14
  Compare the incidence of adverse events between the experimental group and the control group at weeks 2, 6, and 14.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - The Seventh Medical Center, PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Provincial Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - 2nd Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou City Central Hospital, Huzhou, Zhejiang
  - Jinhua City Central Hospital, Jinhua, Zhejiang
  - Quzhou City People's Hospital, Quzhou, Zhejiang
  - The Second Affiliated Hospital, Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No